CLINICAL TRIAL: NCT04623957
Title: Safety and Efficacy of Acupressure Applied Through ForgTin© in Patients With Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pansatori GmbH (Industry)
Collaborators: Competence Center for Medical Devices GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PANSATORI-001
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups whereas both groups will experience the therapy during the course of the clinical investigation.
  Group 1 receives the intervention for a duration of three months. This Phase I is followed by a Washout period of one month and by a non-interventional phase (Phase II).
  Group 2 receives no initial treatment for a duration of three months (Phase I). This Phase I is followed by a Washout period of one month and by an interventional phase (Phase II). Phase III is introduced for both groups for ethical and motivational purposes and to observe potential long-term effects within Group 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ForgTin (Experimental): Patients randomized into group 1 will receive the ForgTin Medical Device for a duration of 3 months.
  Interventions: Device: ForgTin©
- No intervention (No Intervention): Patients randomized into group 2 will receive no device for a duration of 3 months.

INTERVENTIONS:
Device: ForgTin© — The device is clamped behind the ear via two connected temple parts that pressed together around the connecting axis until an individual perfect wearing comfort is achieved. The pressure is adjusted so that the wearing of ForgTin© is barely noticed at all and may be changed at any time.
  The aim is a slight pressure stimulation of clearly defined points behind the ear - thus wearing ForgTin© leads to a minimization of individual tinnitus noises.
  Arms: ForgTin

SUMMARY:
The main objective of this clinical trial is to evaluate the effectiveness and safety of the medical product ForgTin with regard to the impairment and change in the sensation of tinnitus (volume, frequency, psychological stress).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (aged > 18 years)
* Subjective tinnitus in one or both ears with intermittent or continuous symptoms with a duration of > 6 months
* Tinnitus of Grade II, III or IV according to Mini-Tinnitus-Questionnaire (Mini-TF12):

  * Grade II (score of 8-12): moderately distressed
  * Grade III (score of 13-18): severely distressed
  * Grade III (score of 19-24): most severely distressed
* If a drug therapy with psychoactive substances (e.g. antidepressants, anticonvulsants) exists at the beginning of the therapeutic intervention, it must have been stable for at least 30 days. The therapy should remain constant during the duration of the study, but a necessary change is not an exclusion criterion. Any change in medication is documented in the CRF.
* Provides written informed consent

Exclusion Criteria:

* Vestibular schwannoma (acoustic neuroma)
* Objective tinnitus
* Any other tinnitus-related treatment
* Ménière's Disease
* Acute infections of the hearing system (acute otitis media, otitis externa, acute sinusitis)
* Acute infections (acute otitis media, otitis externa, acute sinusitis)
* Hearing aids or Cochlear Implants (CI)
* Any current treatment with anticonvulsants, cortisone, tricyclic antidepressants
* Other lesions (glomus tumors, meningiomas, adenomas, vascular lesions or neuro-vascular conflicts) detected by clinical assessment
* Serious, concomitant disorder, including major depression, anxiety
* Any condition that, in the judgment of the investigator, might prevent safe participation in the study or interfere with study objectives
* Inability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | Change of the Tinnitus Handicap Inventory assessed at Day 0, Month 3, Month 4, Month 7
  Tinnitus Impairment as assessed by the Tinnitus Handicap Inventory (THI)